CLINICAL TRIAL: NCT00550303
Title: An Open-Label, Single-Dose, Non-Randomized, 4-Period Crossover Bioavailability Study of Bazedoxifene Contained in Bazedoxifene/Conjugated Estrogen Tablets Administered to Healthy Postmenopausal Women
Brief Title: Study Comparing Formulations of Bazedoxifene/Conjugated Estrogens
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3115A1-1123
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Healthy
MeSH Terms: interventions — bazedoxifene

INTERVENTIONS:
Drug: bazedoxifene/conjugated estrogens combination

SUMMARY:
The primary purpose is to determine bioavailability of Bazedoxifene/conjugated estrogen formulations for future testing purposes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, post menopausal women ages 45 to 70

Exclusion Criteria:

* Male subjects

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2007-10; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Bioavailability

SECONDARY OUTCOMES:
Safety & tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer